CLINICAL TRIAL: NCT04031248
Title: Effects of the Whole Body Vibration Application and Exercise in Patients With Patellofemoral Pain Syndrome: a Randomized Controlled Trial.
Brief Title: Whole Body Vibration and Exercise in Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: University of Seville (Other)
Responsible Party: Principal Investigator, Sergio Hernandez Sanchez, Lecturer, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0916
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Patello Femoral Syndrome
Keywords: knee; whole body vibration; therapeutic exercise
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WBV group (experimental) (Experimental): Participants in the experimental group will follow a program that will consist of a routine of 18 exercises that will be executed where the greatest neuromuscular recruitment is sought. Most exercises are dynamic and isotonic. It is structured following the scheduled phases (ACSM, 2013) of warm-up, development and return to calm or stretching. The total duration of the program is 22 minutes, keeping the general lines of high-intensity aerobic interval training, which establishes a rest period at least equal to that of work.
  The treatment protocol will consist of 11 sessions applied in 4 weeks under an intervention regime of weeks 3 sessions, with a duration per session of 22 minutes, which will be supervised by a physiotherapist with more than 15 years of clinical experience.
  Interventions: Device: Whole body vibration
- Exercise group (control) (Active Comparator): Control subjects will perform the same exercise program without whole-body vibration.
  Interventions: Other: EXERCISE group

INTERVENTIONS:
Device: Whole body vibration — In this study an axial vibratory platform will be used: POWER-PLATE pro 5 AIRdaptive TM HP®. This device is reviewed annually by the technical unit of the company itself and complies with the international regulations that regulate the Medical Devices [Devices Directive (MDD) 93/42 / EEC (ISO 2631. 2011, Powerplate.com, 2013)]. The vibration will be administered with 2 mm of amplitude and 40 Hz of frequency.
  Arms: WBV group (experimental)
Other: EXERCISE group — The program will consist of a routine of 18 exercises that will be executed where the greatest neuromuscular recruitment is sought. Most exercises are dynamic and isotonic. It is structured following the scheduled phases (ACSM, 2013) of warm-up, development and return to calm or stretching. The total duration of the program is 22 minutes, keeping the general lines of high-intensity aerobic interval training, which establishes a rest period at least equal to that of work. The treatment protocol will consist of 11 sessions applied in 4 weeks under an intervention regime of weeks 3 sessions, with a duration per session of 22 minutes, which will be supervised by a physiotherapist with more than 15 years of clinical experience.
  Arms: Exercise group (control)

SUMMARY:
The present study will consist of evaluating the effect of applying an exercise protocol on a vibratory platform in order to provoke immediate influences in the affected systems and in the quality of life of the patients with patella-femoral pain.

DETAILED DESCRIPTION:
Knee pain is a common condition with a high prevalence in the general population, being femoro-patellar pain one of the most common forms of knee pain (Crossley et al., 2016a). Its incidence ranges between 5.1% and 14.9% and its prevalence is between 16.3% and 28.9% in adolescents (Smith et al., 2018). Femoro-patellar pain is described as diffuse pain in the anterior area of the knee not caused by a traumatic action, which is aggravated when performing squats, running, going up and down stairs or sitting for a long time The recommended conservative treatment for this condition according to the 2016 Manchester and Australia 2017consensus is the therapeutic exercise, combining knee and hip exercises (Crossley et al., 2016b), mainly quadriceps and gluteus medius (Collins et al., 2018).

INTERVENTION All participants will be assessed at baseline and at the end of treatment (discharge) by a blinded investigator.

The program will consist of a routine of 18 exercises that will be executed where the greatest neuromuscular recruitment is sought. Most exercises are dynamic and isotonic. It is structured following the scheduled phases (ACSM, 2013) of warm-up, development and return to calm or stretching. The total duration of the program is 22 minutes, keeping the general lines of high-intensity aerobic interval training, which establishes a rest period at least equal to that of work.

The treatment protocol will consist of 11 sessions applied in 4 weeks under an intervention regime of weeks 3 sessions, with a duration per session of 22 minutes, which will be supervised by a physiotherapist with more than 15 years of clinical experience.

The experimental group will develop the exercise program on the whole body vibration platform, and control group on the switched-off vibration device (without any vibration stimuli)

DESIGN AND STATISTICS

This study will be a randomized clinical trial with a control group. It will consider an alpha or type I error of 95% and a beta or type II error of 80%, with a hypothesis to a tail. The randomized controlled trial will be performed with a single-blind (the evaluator who evaluated the outcome measures remained blinded to the participants' allocation group). The sample will be randomly selected through the randomized.com program among the patients that meet the inclusion criteria that we will be described later. Participants will be distributed equally between the control group and the experimental group.

The research protocol will be carried out in accordance with the Declaration of Helsinki statement of ethics, legal and regulatory principles to provide guidance for research related to health in humans. The CONSORT guidelines have been the reference to design the Project, the ad will be used to make the final report.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with pain in the anterior aspect of the knee.
* Participants with a self-reported pain intensity ≥ 30 mm on the Visual Analogue Scale

Exclusion Criteria:

* any contraindication for the use of training with whole-body vibration;
* to have received knee injections of corticosteroids or hyaluronic acid;
* cognition or impaired communication;
* to be involved in an ongoing medical-legal dispute.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Visual Analog Scale (VAS). For the assessment of pain intensity during activity we will use an analogue scale of 10 centimeters, in which, 0 corresponds to "no pain" and 10 represents the "worst pain imaginable". The VAS of 10 centimeters is trusted and validated.
  The questionnaire Douleur Neuropathique-4 items (DN4) (Bouhassira D, et al., 2005).
  In order to assess neuropathic pain, we have used the Spanish validated version of the DN4 (Perez et al., 2007). This questionnaire consists of 10 items, consisting of descriptions and signs of pain that are evaluated with 1 (yes) or 0 (no) that indicate patients who have a high probability of having a neuropathic pain component. The evaluations of the individual items are added to obtain a maximum total score of 10, with a cut-off point ≥4.
Pain intensity | After treatment (Discharge, 4 weeks)
  Visual Analog Scale (VAS). For the assessment of pain intensity during activity we will use an analogue scale of 10 centimeters, in which, 0 corresponds to "no pain" and 10 represents the "worst pain imaginable". The VAS of 10 centimeters is trusted and validated.
  The questionnaire Douleur Neuropathique-4 items (DN4) (Bouhassira D, et al., 2005).
  In order to assess neuropathic pain, we have used the Spanish validated version of the DN4 (Perez et al., 2007). This questionnaire consists of 10 items, consisting of descriptions and signs of pain that are evaluated with 1 (yes) or 0 (no) that indicate patients who have a high probability of having a neuropathic pain component. The evaluations of the individual items are added to obtain a maximum total score of 10, with a cut-off point ≥4.

SECONDARY OUTCOMES:
Knee range of movement | Baseline
  Goniometer (Norkin, 1997; Hancock et al., 2018). Knee flexion ROM measurement The individual was placed at dorsal decubitus, with 90 degrees of hip flexion. Hip positioning was guaranteed by the use of a thigh device which aided in the maintenance of the pre-set position. The universal goniometer was placed next to the femoral lateral epicondyle. The static handle of the goniometer was aligned with the thigh, having the femoral major trochanter as reference and the mobile handle aligned with the leg, with reference in the fibula lateral malleolus. The digital inclinometer was placed proximal and anteriorly on the leg, resting on the tibial crest.
  Knee extension ROM measurement The individual was at dorsal decubitus, with extended legs. The evaluated limb was raised by the heel, with knee stabilization in contact with the stretcher. The instruments positioning in relation to the segment was the same of the measurements performed for knee flexion.
Knee range of movement | After treatment (Discharge, 4 weeks)
  Goniometer (Norkin, 1997; Hancock et al., 2018). Knee flexion ROM measurement The individual was placed at dorsal decubitus, with 90 degrees of hip flexion. Hip positioning was guaranteed by the use of a thigh device which aided in the maintenance of the pre-set position. The universal goniometer was placed next to the femoral lateral epicondyle. The static handle of the goniometer was aligned with the thigh, having the femoral major trochanter as reference and the mobile handle aligned with the leg, with reference in the fibula lateral malleolus. The digital inclinometer was placed proximal and anteriorly on the leg, resting on the tibial crest.
  Knee extension ROM measurement The individual was at dorsal decubitus, with extended legs. The evaluated limb was raised by the heel, with knee stabilization in contact with the stretcher. The instruments positioning in relation to the segment was the same of the measurements performed for knee flexion.
Disability and functional assessment | Baseline
  Functional Scale of the Lower Extremity (LEFS). The Spanish version of this self-report questionnaire will be applied. This scale consists of 20 items with a score of 0 to 4, where the highest score represents the highest functionality of the lower limb (Cruz-Díaz et al., 2014, Binkley et al., 1999).
  Kujala Patellofemoral Score. We will use the validated Spanish version of the validated questionnaire of 13 items, which designate a specific self-report of how each subject with patello.femoral pain perceives the function of the knee. Each item is based on six points where the highest scores represent a better functional capacity (Corum et al., 2018, Martínez-cano et al., 2017)
Disability and functional assessment | After treatment (Discharge, 4 weeks)
  Functional Scale of the Lower Extremity (LEFS). The Spanish version of this self-report questionnaire will be applied. This scale consists of 20 items with a score of 0 to 4, where the highest score represents the highest functionality of the lower limb (Cruz-Díaz et al., 2014, Binkley et al., 1999).
  Kujala Patellofemoral Score. We will use the validated Spanish version of the validated questionnaire of 13 items, which designate a specific self-report of how each subject with patello.femoral pain perceives the function of the knee. Each item is based on six points where the highest scores represent a better functional capacity (Corum et al., 2018, Martínez-cano et al., 2017)

CONTACTS AND LOCATIONS:
Locations (1):
- A360 Heath and Sport Clinic, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yanez-Alvarez A, Bermudez-Pulgarin B, Hernandez-Sanchez S, Albornoz-Cabello M. Effects of exercise combined with whole body vibration in patients with patellofemoral pain syndrome: a randomised-controlled clinical trial. BMC Musculoskelet Disord. 2020 Aug 28;21(1):582. doi: 10.1186/s12891-020-03599-2. PMID 32859183